CLINICAL TRIAL: NCT03505437
Title: The Impact of Stress on Exposure-based Treatment Outcome
Brief Title: Effects of Stress on Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Armin Zlomuzica, Dr. / Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FP 1-2
Record Dates: First submitted 2018-02-01; First posted 2018-04-23 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Specific Phobia
Keywords: anxiety disorders; spider phobia; stress; exposure therapy; generalization
MeSH Terms: conditions — Phobia, Specific; Anxiety Disorders; Arachnophobia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress + Exposure (Experimental): Stress Condition: Cold water condition of the socially evaluated cold pressor test (SECPT; Schwabe et al, 2008).
  Interventions: Other: Cold water condition
- Control + Exposure (Active Comparator): Control condition: Warm water condition of the SECPT.
  Interventions: Other: Warm water condition

INTERVENTIONS:
Other: Cold water condition — Cold water condition of the SECPT. Participants immerse their hand into ice-cold water (0-3°C). During the SECPT, participants are videotyped and monitored. After the SECPT, participants will receive 45 minutes of in-vivo exposure to spiders
  Arms: Stress + Exposure
Other: Warm water condition — Warm water condition of the SECPT. Participants immerse their hand into warm water (36-37°C). Participants are neither videotyped nor monitored during the whole procedure. After the SECPT, participants will receive 45 minutes of in-vivo exposure to spiders.
  Arms: Control + Exposure

SUMMARY:
This study investigates whether stress can augment exposure therapy outcome in patients with specific phobia (spider phobia).

DETAILED DESCRIPTION:
Stress has been shown to modulate fear extinction. The present study is aimed at investigating whether stress (administered prior to exposure with the socially evaluated cold pressor test) augments exposure therapy outcome in patients with specific phobia (spider phobia). Furthermore, the effects of stress on the generalization of exposure-induced symptom reduction towards untreated fear stimuli (i.e. cockroaches) will be explored.

Participants are randomly assigned to the cold or warm water condition of the socially evaluated cold pressor test (SECPT; Schwabe et al., 2008). Thereafter, participants of both conditions receive 45 minutes of in-vivo exposure to spiders. The effects of stress on exposure-based anxiety reductions toward spiders (treated fear stimulus) and cockroaches (untreated fear stimulus to assess generalization of treatment outcome) are assessed on the behavioral, subjective and physiological level at pretreatment, posttreatment (24 hours after exposure) and follow-up (4 weeks after exposure).

ELIGIBILITY:
Inclusion Criteria:

* Women using oral contraceptives (OC)
* Specific phobia (spider phobia)

Exclusion Criteria:

* Body Mass Index (BMI) < 19 or > 27
* Pregnancy
* Any acute or chronic mental, somatic, endocrine, or metabolic disease
* Psychological, psychiatric, neurological or pharmacological treatment
* Shift work
* Smoking more than 5 cigarettes per month
* Vaccination in the past 2 month
* Drug or alcohol abuse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in the Behavioral Approach Test (BAT) with spiders (treated fear stimulus) | Pretreatment, Posttreatment, Follow-up (with approx. 1 day between pre- and posttreatment and 4 weeks between pretreatment and follow-up)
  During the Behavioral Approach Test (BAT) the closest distance to a spider as well as subjective fear and heart rate is measured.
Change in the Behavioral Approach Test with Cockroaches (untreated fear stimulus) | Pretreatment, Follow-up (with approx. 4 weeks between pretreatment and follow-up)
  During the Behavioral Approach Test (BAT) the closest distance to a cockroach as well as subjective fear and heart rate is measured.

SECONDARY OUTCOMES:
Change in the Spider-fear Related questionnaires | Pretreatment, Posttreatment, Follow-up (with approx. 1 day between pre- and posttreatment and 4 weeks between pretreatment and follow-up)
  Self-report questionnaires assessing fear of spiders will be used. The Fear of Spiders Questionnaire (FSQ) and the Spider Beliefs Questionnaire (SBQ) will be employed. Scores on these scales range from 0 to 108 and 0 to 100, respectively, with higher scores indicating greater fear of spiders.
Change in the Cockroach-fear related questionnaires | Pretreatment, Posttreatment, Follow-up (with approx. 1 day between pre- and posttreatment and 4 weeks between pretreatment and follow-up)
  Self-report questionnaires assessing fear of cockroaches will be used. The Fear of Cockroach Questionnaire and the Cockroach Beliefs Questionnaire will be employed. Scores on these scales range from 0 to 108 and 0 to 100, respectively, with higher scores indicating greater fear of cockroaches.
Free cortisol concentrations | 5 times at Pretreatment, 2 times at Posttreatment, 2 times at Follow-up. (with approx. 1 day between pre- and posttreatment and 4 weeks between pretreatment and follow-up)
  Manipulation check (SECPT). Saliva will be collected using salivette sampling devices (Sarstedt, Nümbrecht) at different time points to assess free cortisol concentrations and activity of the enzyme alpha amylase
Blood pressure | 9 times at Pretreatment
  Manipulation check (SECPT). Systolic and diastolic blood pressure (mm/Hg) are measured at different time points
Activity of the enzyme alpha amylase | 5 times at Pretreatment, 2 times at Posttreatment, 2 times at Follow-up ( (with approx. 1 day between pre- and posttreatment and 4 weeks between pretreatment and follow-up)
  Alpha amylase will be collected using salivette sampling devices

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zlomuzica, PhD, Principal Investigator — Ruhr-University Bochum
Locations (1):
- Mental Health Research and Treatment Center, Bochum, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwabe L, Haddad L, Schachinger H. HPA axis activation by a socially evaluated cold-pressor test. Psychoneuroendocrinology. 2008 Jul;33(6):890-5. doi: 10.1016/j.psyneuen.2008.03.001. Epub 2008 Apr 9. PMID 18403130